CLINICAL TRIAL: NCT03957161
Title: Angiotensin-converting Enzyme Inhibitors (ACEi) or Angiotensin Receptor Blockers (ARB) Withdrawal in Patients With Advanced Chronic Kidney Disease
Brief Title: ACEi ARB Withdrawal in CKD Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Currently we are not pursuing this trial due t o limited bandwidth and have not enrolled any participants.
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-25554
Record Dates: First submitted 2019-05-15; First posted 2019-05-21 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Chronic Kidney Disease; Blood Pressure; Angiotensin-converting Enzyme Inhibitor; Angiotensin Receptor Blockers
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACEi/ARB continuation (Experimental): Intervention group will continue or start to take ACEi and/or ARBs
  Interventions: Other: Continuation of ACEi and/or ARBs
- ACEi/ARB withdrawal (No Intervention): The control group will discontinue ACEi and/or ARBs which may be substituted with other anti-hypertensive agents (if already taking ACEi/ARB) or continue to not take ACEi/ARBs

INTERVENTIONS:
Other: Continuation of ACEi and/or ARBs — Patients will continue or start taking ACEi and/or ARBs
  Arms: ACEi/ARB continuation

SUMMARY:
The American Heart Association guidelines for high blood pressure (BP) currently recommend using angiotensin-converting enzyme inhibitors (ACEi) or angiotensin receptor blockers (ARBs) as first-line therapy for patients with chronic kidney disease (CKD) stage 3 or above. However, the prevalence of ACEi and ARB use in patients with CKD stage 4 or 5 is low, and current BP guidelines acknowledge the lack of solid evidence to support the benefit of using these agents in advanced CKD.This study seeks to conduct a pilot trial to determine the safety and feasibility of ACEi and/or ARB continuation (intervention) versus withdrawal (control) in patients with advanced CKD.

ELIGIBILITY:
Inclusion Criteria:

* adults ≥18 years of age who meet the eGFR eligibility criteria, which will be determined based on whether participants have at least two eGFR in the last three months that are < 25 mL/min/1.73m2 or prior diagnosis of CKD (per electronic chart review) and at least one eGFR < 25 mL/min/1.73m2 in the past six months
* receiving at least one antihypertensive medication at the time of the screening visit.

Exclusion Criteria:

The investigators will exclude those who:

* are or are planning to become pregnant, due to inability to take multiple classes of anti-hypertensive agents
* are marginally housed, due to concerns regarding routine follow-up
* are actively participating in a different interventional trial that may affect blood pressure
* are unwilling to consent to participate
* institutionalized individuals or prisoners
* are actively abusing illicit drugs or alcohol
* have a history of poor or doubtful compliance (e.g., frequently missed appointments)
* have cognitive impairment prohibiting participation in the study
* on dialysis at time of recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Rate of enrollment and dropout in trial | Months 1-12
  measure of acceptability of continuing ACEi/ARBs among providers and patients
Number of patients who have onset of hyperkalemia (non-hemolyzed potassium ≥6.0 meq/L) | Months 1-12
  safety measure
Number of all cause emergency room visits | Months 1-12
  safety measure
Number of all-cause hospitalizations | Months 1-12
  safety measure
Number of falls and syncope reported by patients and/or discharge summaries | Months 1-12
  safety measure
Number of patients who receive chronic dialysis or kidney transplant | Months 1-12
  Marks the onset of end-stage renal disease

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Ku, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No